CLINICAL TRIAL: NCT02694536
Title: A Phase IIIb Study of Tarceva (Erlotinib) in Patients With Locally Advanced, Unresectable or Metastatic Pancreatic Cancer
Brief Title: A Study of Erlotinib in Locally Advanced, Unresectable, or Metastatic Pancreatic Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ML19537; 2005-004605-29 (EudraCT Number)
Record Dates: First submitted 2016-02-24; First posted 2016-02-29 (Estimated); Results first posted 2017-01-10 (Estimated); Last update posted 2017-03-24 (Actual); Status verified 2017-02

CONDITIONS: Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Erlotinib Hydrochloride; Gemcitabine

ARMS (1):
- Erlotinib + Gemcitabine (Experimental): Participants will receive erlotinib in combination with standard of care chemotherapy (gemcitabine) until disease progression, unacceptable toxicity, or withdrawal for any reason.
  Interventions: Drug: Erlotinib; Drug: Gemcitabine

INTERVENTIONS:
Drug: Erlotinib — Participants will receive erlotinib tablets as 100 milligrams (mg) orally (PO) once daily.
  Other Names: Tarceva
Drug: Gemcitabine — Participants will receive gemcitabine as 1000 milligrams per meter-squared (mg/m^2) via intravenous (IV) infusion on Days 1, 8, 15, 22, 29, 36, and 43 of the first 8-week cycle, and thereafter on Days 1, 8, and 15 of every 4-week cycle.

SUMMARY:
This open-label, single-arm, multicenter trial is designed to evaluate the safety of erlotinib in combination with standard of care chemotherapy (gemcitabine) in participants with locally advanced, unresectable, or metastatic pancreatic cancer.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed adenocarcinoma with locally advanced, unresectable, or metastatic disease
* No prior systemic treatment for metastatic disease
* Adjuvant therapy ≥6 months prior to study entry with no residual toxic effects
* Eastern Cooperative Oncology Group (ECOG) performance status 0 to 3
* Life expectancy ≥12 weeks
* Adequate hematologic, hepatic, and renal function
* Negative pregnancy test within 72 hours of study drug and use of effective contraception among women of childbearing potential

Exclusion Criteria:

* Unstable systemic disease
* Prior systemic human epidermal growth factor receptor 1 (HER1) or epidermal growth factor receptor (EGFR) inhibitors
* Other malignancy within 5 years prior to study entry
* Significant opthalmologic abnormality
* Inability to take oral medication
* Need for IV alimentation
* Prior surgery affecting absorption
* Active peptic ulcer disease
* Nursing mothers

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2006-08-01; Primary Completion 2009-11-19 (Actual); Study Completion 2009-11-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Chair — Hoffmann-La Roche
Locations (11):
- Italy (11):
  - Bari, Apulia
  - Napoli, Campania
  - Bologna, Emilia-Romagna
  - Pordenone, Friuli Venezia Giulia
  - Rome, Lazio
  - Pavia, Lombardy
  - Catania, Sicily
  - Pisa, Tuscany
  - Perugia, Umbria
  - Cona (Ferrara), Veneto
  - Verona, Veneto

RESULTS

PARTICIPANT FLOW:
Groups:
- Erlotinib + Gemcitabine: Participants with locally advanced, unresectable, or metastatic pancreatic cancer received erlotinib in combination with standard of care chemotherapy (gemcitabine) until disease progression, unacceptable toxicity, or withdrawal for any reason. Erlotinib was administered as 100 milligrams (mg) orally (PO) once daily. Gemcitabine was administered as 1000 milligrams per meter-squared (mg/m^2) via intravenous (IV) infusion on Days 1, 8, 15, 22, 29, 36, and 43 of the first 8-week cycle, and thereafter on Days 1, 8, and 15 of every 4-week cycle.
Period: Overall Study
Arm/Group | Erlotinib + Gemcitabine
Started | 80
Completed | 0
Not Completed | 80
Not completed — Progressive Disease | 40
Not completed — Lost to Follow-up | 1
Not completed — Study Drug-Related Adverse Event | 1
Not completed — Withdrawal by Subject | 8
Not completed — Death | 8
Not completed — Other | 22

BASELINE CHARACTERISTICS:
Population: Safety Population: All participants who received at least one dose of erlotinib.
Groups:
- Erlotinib + Gemcitabine: Participants with locally advanced, unresectable, or metastatic pancreatic cancer received erlotinib in combination with standard of care chemotherapy (gemcitabine) until disease progression, unacceptable toxicity, or withdrawal for any reason. Erlotinib was administered as 100 mg PO once daily. Gemcitabine was administered as 1000 mg/m^2 via IV infusion on Days 1, 8, 15, 22, 29, 36, and 43 of the first 8-week cycle, and thereafter on Days 1, 8, and 15 of every 4-week cycle.
Arm/Group | Erlotinib + Gemcitabine
Number analyzed (Participants) | 80
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.45 (10.299)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32
  Male | 48

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Adverse Events (AEs)
Description: An AE was defined as any untoward medical occurrence and which did not necessarily have a causal relationship with treatment. The percentage of participants who experienced at least 1 AE was reported.
Time Frame: Up to approximately 40 months (assessed continuously during treatment)
Population: Safety Population
Measure: Number; unit: percentage of participants
Arm/Group | Erlotinib + Gemcitabine
Number analyzed (Participants) | 80
percentage of participants | 78.8

2. Secondary Outcome: European Organisation for Research and Treatment of Cancer (EORTC) 30-Item Quality of Life Questionnaire (QLQ-C30) Item Scores
Description: The QLQ-C30 is a 30-item questionnaire that assesses physical (Questions 1-5), role (Questions 6-7), emotional (Questions 21-24), cognitive (Questions 20 and 25), and social (Questions 26-27) functional domains as well as global health status (Questions 29-30) and several symptoms including fatigue (Questions 10, 12, and 18), pain (Questions 9 and 19), nausea/vomiting (Questions 14-15), dyspnea (Question 8), appetite loss (Question 13), insomnia (Question 11), constipation/diarrhea (Questions 16-17), and financial difficulties (Question 28). Questions 1 to 28 were assessed on a 4-point scale from 1 ("no/not at all") to 4 ("very much") where higher scores represented worse symptoms. Questions 29 and 30 were assessed on a 7-point scale from 1 ("very poor") to 7 ("excellent") where higher scores represented better functioning. Item scores over the study period were averaged among all participants across all visits for which data were available.
Time Frame: Up to approximately 40 months (assessed at Baseline, every 4 weeks during treatment, and end of study)
Population: Safety Population. The "Number of Participants Analyzed" reflects the total number of participants who contributed to the endpoint. The number of responses for each questionnaire item combined across all assessments (n) is shown in the table.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Erlotinib + Gemcitabine
Number analyzed (Participants) | 80
units on a scale
  Q1: Trouble in strenuous activities (n=256) | 1.96 (0.758)
  Q2: Trouble with long walk (n=259) | 2.03 (0.802)
  Q3: Trouble with short walk (n=258) | 1.50 (0.696)
  Q4: Need to say in bed or chair (n=255) | 1.87 (0.699)
  Q5: Need help in daily activities (n=259) | 1.21 (0.501)
  Q6: Limited in doing work/daily activities (n=257) | 1.82 (0.803)
  Q7: Limited in pursuing hobbies (n=255) | 1.73 (0.798)
  Q8: Short of breath (n=258) | 1.38 (0.608)
  Q9: Pain (n=257) | 1.88 (0.771)
  Q10: Need to rest (n=255) | 2.05 (0.697)
  Q11: Trouble sleeping (n=257) | 1.74 (0.699)
  Q12: Felt weak (n=255) | 2.05 (0.774)
  Q13: Lacked appetite (n=257) | 1.70 (0.730)
  Q14: Felt nauseated (n=257) | 1.48 (0.679)
  Q15: Vomited (n=259) | 1.10 (0.414)
  Q16: Constipated (n=259) | 1.51 (0.723)
  Q17: Diarrhea (n=259) | 1.27 (0.496)
  Q18: Tired (n=255) | 2.07 (0.689)
  Q19: Pain interference with daily activity (n=256) | 1.69 (0.814)
  Q20: Difficulty concentrating (n=257) | 1.49 (0.638)
  Q21: Felt tense (n=256) | 1.97 (0.716)
  Q22: Worried (n=253) | 2.10 (0.773)
  Q23: Felt irritable (n=258) | 1.75 (0.707)
  Q24: Felt depressed (n=258) | 1.67 (0.658)
  Q25: Difficulty remembering things (n=257) | 1.44 (0.543)
  Q26: Interference with family life (n=257) | 1.59 (0.680)
  Q27: Interference with social activities (n=257) | 1.62 (0.772)
  Q28: Financial difficulties (n=258) | 1.32 (0.655)
  Q29: Overall health (n=255) | 4.44 (1.314)
  Q30: Overall quality of life (n=255) | 4.38 (1.346)

3. Secondary Outcome: Percentage of Participants Who Died
Description: The percentage of participants who died from any cause was reported to the nearest integer.
Time Frame: Up to approximately 40 months (assessed continuously through end of study)
Population: Safety Population. The "Number of Participants Analyzed" reflects the number of participants who contributed to the endpoint.
Measure: Number; unit: percentage of participants
Arm/Group | Erlotinib + Gemcitabine
Number analyzed (Participants) | 78
percentage of participants | 73

4. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the time from start of treatment to time of death from any cause. Participants who had not died at the time of final analysis were censored at the date of last contact. OS was estimated by Kaplan-Meier methodology and expressed in months.
Time Frame: Up to approximately 40 months (assessed continuously through end of study)
Population: as for outcome 3
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Erlotinib + Gemcitabine
Number analyzed (Participants) | 78
months | 7.49 [5.42 to 9.04]

5. Secondary Outcome: Percentage of Participants With Death or Disease Progression According to Response Evaluation Criteria in Solid Tumors (RECIST)
Description: Tumor assessments were performed using RECIST. Disease progression was defined as greater than or equal to (≥) 20 percent (%) increase in sum of longest diameters (LD) of target lesions in reference to smallest sum of LD on study. The percentage of participants who died or demonstrated disease progression was reported to the nearest integer.
Time Frame: Up to approximately 40 months (assessed at Baseline, every 8 weeks during treatment, and end of study)
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Erlotinib + Gemcitabine
Number analyzed (Participants) | 78
percentage of participants | 88

6. Secondary Outcome: Progression-Free Survival (PFS) According to RECIST
Description: Tumor assessments were performed using RECIST. PFS was defined as the time from treatment start to the time of death or disease progression. Disease progression was defined as ≥20% increase in sum of LD of target lesions in reference to smallest sum of LD on study. PFS was estimated by Kaplan-Meier methodology and expressed in months.
Time Frame: Up to approximately 40 months (assessed at Baseline, every 8 weeks during treatment, and end of study)
Population: as for outcome 3
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Erlotinib + Gemcitabine
Number analyzed (Participants) | 78
months | 4.864 [3.484 to 5.850]

ADVERSE EVENTS:
Time Frame: Up to approximately 40 months (assessed continuously during treatment)
Description: Analysis Population Description: Safety Population.
Arm/Group | Erlotinib + Gemcitabine
Serious Adverse Events (participants affected / at risk) | 35/80
Other Adverse Events (participants affected / at risk) | 44/80
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Erlotinib + Gemcitabine (N=80)
Anaemia (Blood and lymphatic system disorders) | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1
Cardiac arrest (Cardiac disorders) | 2
Myocardial infarction (Cardiac disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 3
Intestinal obstruction (Gastrointestinal disorders) | 1
Intestinal perforation (Gastrointestinal disorders) | 1
Pancreatic carcinoma (Gastrointestinal disorders) | 2
Peritonitis (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Disease progression (General disorders) | 6
General physical health deterioration (General disorders) | 2
Ill-defined disorder (General disorders) | 1
Pyrexia (General disorders) | 1
Hepatic failure (Hepatobiliary disorders) | 2
Jaundice (Hepatobiliary disorders) | 3
Liver abscess (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 2
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3
Cerebrovascular accident (Nervous system disorders) | 2
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1
Surgery (Surgical and medical procedures) | 1
Deep vein thrombosis (Vascular disorders) | 1
Melaena (Blood and lymphatic system disorders) | 1
Ileus (Gastrointestinal disorders) | 1
Multi-organ failure (General disorders) | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Erlotinib + Gemcitabine (N=80)
Anaemia (Blood and lymphatic system disorders) | 21
Thrombocytopenia (Blood and lymphatic system disorders) | 18
Leukopenia (Blood and lymphatic system disorders) | 14
Neutropenia (Blood and lymphatic system disorders) | 9
Constipation (Gastrointestinal disorders) | 5
Abdominal pain (Gastrointestinal disorders) | 4
Pyrexia (General disorders) | 12
Asthenia (General disorders) | 4
Hepatotoxicity (Hepatobiliary disorders) | 5
Alanine aminotransferase increased (Investigations) | 5
Aspartate aminotransferase increased (Investigations) | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.